CLINICAL TRIAL: NCT07272720
Title: Post-Market Clinical Follow-Up Investigation of MODULITH® SLX-F2 With StorM-Track in Patients With Kidney Stones - A Confirmatory Parallel-Group, Randomized Controlled Trial
Brief Title: PMCF Investigation of MODULITH® SLX-F2 With StorM-Track in Patients With Kidney Stones
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Storz Medical AG (Industry)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIV-25-05-052934
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Kidney Stones; Urolithiasis
Keywords: Kidney stones; Urolithiasis; Extracorporeal shockwave lithotripsy; ESWL
MeSH Terms: conditions — Kidney Calculi; Urolithiasis | interventions — Lithotripsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWL with kidney stone tracking (StorM-Track). (Experimental)
  Interventions: Device: ESWL with kidney stone tracking (StorM-Track)
- Standard ESWL without stone tracking (StorM-Track disabled). (Active Comparator)
  Interventions: Device: Standard ESWL without stone tracking (StorM-Track disabled)

INTERVENTIONS:
Device: ESWL with kidney stone tracking (StorM-Track) — Starting ESWL on a low energy setting with stepwise ramping and at a frequency of 1.0 or 1.5 Hz.
  Up to a maximum of 3'500 shockwaves unless there is no stone visible in X-ray imaging.
  If fragments > 4mm remain after the first ESWL treatment, a 2nd ESWL will be performed.
  Arms: ESWL with kidney stone tracking (StorM-Track).
Device: Standard ESWL without stone tracking (StorM-Track disabled) — Same treatment protocol as for the intervention group.
  If fragments > 4mm remain after the first ESWL treatment, a 2nd ESWL will be performed.
  Arms: Standard ESWL without stone tracking (StorM-Track disabled).

SUMMARY:
Extracorporeal shockwave lithotripsy (ESWL) is a non-invasive standard treatment for kidney stones.

This study will be conducted to evaluate the effectiveness of ESWL using MODULITH® SLX-F2 with stone tracking, compared to MODULITH® SLX-F2 without stone tracking, in adult patients with kidney stones, as measured by stone-free status.

DETAILED DESCRIPTION:
The success of ESWL depends on multiple procedure- and patient-specific factors, one crucial factor being accurate stone targeting. Respiration induced kidney movement affects stone targeting as it results in the stone not being hit by the shock waves for up to 50% of the treatment time.

To improve the accuracy of stone targeting and comminution, an additional tracking module has been incorporated into the state-of-the-art lithotripter MODULITH® SLX-F2. The device is CE marked including its tracking module.

The scientific rationale for conducting this clinical investigation is based on the hypothesis that improved stone targeting through real-time tracking may lead to increased treatment efficacy and safety, as reflected by higher stone-free rates, reduced need for re-treatment, an increased quality of life, and lower adverse events rates.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Single kidney stone (6 - 15 mm) in the target kidney
3. Stone density assessed by Hounsfield unit value (HU) ≤ 1,200 HU

Exclusion Criteria:

1. BMI > 29.9
2. Target stone that cannot be localised
3. Multiple kidney stones in the target kidney
4. Stones with a density value of > 1,200 HU
5. Skin to stone distance (SSD) > 160 mm
6. The presence of obstructions, malformations or other factors preventing targeting or passing of the stone, including but not limited to the following:

   1. Skeletal malformations and obesity, preventing targeting of the stone
   2. Malignant tumour in the shockwave path
   3. Arterial aneurysm or calcium deposits, or thrombosis in shockwave path
   4. Brain, spinal column or air-filled tissue, especially the lungs, in the shockwave path
   5. Obstruction distal to the stone (as this would hinder the passage of fragments through collecting system or ureter)
7. Any disease/medical condition, prior or concomitant medication/treatment/intervention, or implant that may affect this clinical investigation, and/or is contraindicated for the IMD, including but not limited to the following:

   1. Severe nephrocalcinosis
   2. Uncontrolled urinary tract infection
   3. Coagulation disorders and bleeding diathesis, not compensated according to urological and hemostaseological guidelines
   4. Anticoagulation or platelet inhibition therapy, not bridged according to urological and hemostaseological guidelines
   5. Uncontrolled hypertension
   6. Blood pressure > 180/100
   7. Active cardiac implants that are not authorized for use with ESWL
   8. Pancreatitis
   9. Ehlers-Danlos syndrome
   10. Administration of contrast agents containing gases for ultrasound diagnostics less than 24 hours before treatment.
8. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Stone-free rate (SFR) | 6±2 weeks post 1st treatment
  Proportion of subjects who are stone free or present with clinically insignificant residual fragments (measuring ≤ 4 mm on CT)

OTHER OUTCOMES:
Stone free rate (SFR) | 12±4 weeks post 1st treatment
  Proportion of subjects who are stone free or present with clinically insignificant residual fragments (measuring ≤ 4 mm on CT).
  Only for subjects who had a 2nd ESWL treatment at 6±2 weeks.
Stone free rate | 12±1 months post 1st treatment
  Proportion of subjects who are stone free or present with clinically insignificant residual fragments (measuring ≤ 4 mm on CT)
Proportions of subjects with stone-free status classified into grades | 6±2 weeks post 1st treatment
  Grade A (completely stone free, no stones on CT scan); Grade B (Grade A stones plus ≤ 2 mm fragments); Grade C (Grade A and B stones plus C 2.1 - 4 mm fragments)
Proportions of subjects with stone-free status classified into grades | 12±4 weeks post 1st treatment
  Grade A (completely stone free, no stones on CT scan); Grade B (Grade A stones plus ≤ 2 mm fragments); Grade C (Grade A and B stones plus C 2.1 - 4 mm fragments).
  Only for subjects who had a 2nd ESWL treatment at 6±2 weeks.
Proportions of subjects with stone-free status classified into grades | 12±1 months post 1st treatment
  Grade A (completely stone free, no stones on CT scan); Grade B (Grade A stones plus ≤ 2 mm fragments); Grade C (Grade A and B stones plus C 2.1 - 4 mm fragments)
Change from baseline in the mean total WISQOL score | Baseline, 6±2 weeks post 1st treatment
  Wisconsin Stone Quality of Life Questionnaire (WISQOL).
  WISQOLTotal "raw" score = min-max 28-140 (lowest to highest QOL).
  WISQOLTotal "standardized" score = min-max 0-100 (lowest to highest QOL).
ESWL re-treatment rate | 12±1 months post 1st treatment
  The proportion of subjects with a need for re-treatment with ESWL during the 12 months follow-up period.
Auxiliary procedures rate | 12±1 months post 1st treatment
  The proportion of subjects with need for auxiliary procedures during the 12 months follow-up period.
Duration of hospital stay | 12±1 months post 1st treatment
  The total number of days in hospital per subject
Total adverse device effect (ADE) rate | 6±2 weeks post 1st treatment
  The number of ADEs (mild, moderate, severe; CTCAE v5.0 or higher) divided by the number of subjects.
Total adverse device effect (ADE) rate | 12±4 weeks post 1st treatment
  The number of ADEs (mild, moderate, severe; CTCAE v5.0 or higher) divided by the number of subjects.
  Only for subjects who had a 2nd ESWL treatment.
Total adverse device effect (ADE) rate | 12±1 months post 1st treatment
  The number of ADEs (mild, moderate, severe; CTCAE v5.0 or higher) divided by the number of subjects
Adverse device effect (ADE) incidence | 6±2 weeks post 1st treatment
  the number of subjects with one or more ADE (mild, moderate, severe; CTCAE v5.0 or higher)
Adverse device effect (ADE) incidence | 12±4 weeks post 1st treatment
  The number of subjects with one or more ADE (mild, moderate, severe; CTCAE v5.0 or higher).
  Only for subjects who had a 2nd ESWL treatment.
Adverse device effect (ADE) incidence | 12±1 months post 1st treatment
  The number of subjects with one or more ADE (mild, moderate, severe; CTCAE v5.0 or higher).
Mean total radiation dose area product (DAP) [μGy·m²] per subject | 12±1 months post 1st treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No